CLINICAL TRIAL: NCT04197544
Title: Evaluation of the Implantation of the End-vascular Creation of the Arteriovenous Fistulas in Patients in the University Hospital of Araba. Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fernando López Zárraga (Other Government)
Responsible Party: Sponsor-Investigator, Fernando López Zárraga, Principal Investigator, Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAVIS
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Efficacy and Safety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Procedure: endoFAVI
- Control group (No Intervention)

INTERVENTIONS:
Procedure: endoFAVI — EndoFAVI creation to patients that require vascular access for hemodialysis.
  Arms: Intervention group

SUMMARY:
In last few years, there is a new technology that permits the endovascular fistula creation with a minimum vascular trauma and the first results show encouraging results with high technical success rate, low resurgent and failure rates and good usability for hemodialysis.

The implementation of the endoFAVI realization in dialysis patients is an emergent procedure that in our hospital can contribute important benefits to the patients, savings to the health system, as well research and innovation in the implicate services.

ELIGIBILITY:
Inclusion Criteria:

* Adult (older than 18).
* Currently be receiving chronic dialysis, or be waiting to start the chronic dialysis in the next six months.
* Have veins with diameter >= 2.0mm to the creation of the fistula, established by Duplex ultrasound or venogram.
* Have arteries with diameter >= 2.0mm to the creation of the fistula, established by Duplex ultrasound or venogram.
* Cubital and radial arterial flow for the hand, confirmed with Duplex Ultrasound and/or Allen test.
* Dismissed the realization of cephalic-radius FAVI for surgical technical problems.
* Informed Consent to participate in the study.

Exclusion Criteria:

* Known central venous stenosis or narrowing of the central vein > 50% according to images on the same side as the creation of the planned FAV.
* Absence of perforator that feed the target cannulation, by venogram.
* Occlusion or stenosis > 50% of the cephalic basilica vein of the target cannulation.
* Cannulation target vein of less than 2.0 mm of diameter.
* Significantly compromised flow (>= 50% of stenosis) in the treatment arm as determined by the doctor and the images.
* Ejection fraction documented <= 35% in the last 6 months.
* Pregnant women.
* Heart failure Class III or IV of the New York Heart Association (NYHA).
* Hypercouagulability status demonstrated ( Antiphospholipid Syndrome, Leiden factor V, Protein deficit S, ...).
* Known hemorrhagic diathesis.
* Documented history of drug abuse including intravenous drugs within six months of FAV creation.
* Concomitant major surgical procedure "planned" within three months of recruitment or major previous surgery within 30 days of recruitment.
* Known iodine contrast allergy that cannot be properly premedicated.
* Known adverse effects for sedation and/or anesthesia that cannot be properly premedicated.
* Evidence of active infections on the day of the index procedure.
* Life expectancy < 1 year.
* The patient is not willing to provide an written informed consent, is not geographically stable and/or is not willing to cmply with the required follow-up.
* Patient with an objective cannulation vein of more than 6 mm of deep that would require a transposition procedure, defined as the elevation of an objective cannulation vein nad the creation of a new fistula AV.
* The patient is nit willing to undergo of second stage, defined as a conversion to surgical FAVI, central catheter arrangement, thrombectomy/rescue fibrinolysis, stenoic area angioplasty, ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of endoFAVI physiologically appropriate for the hemodialysis during the next three months to the creation. | Three months next the creation
  The absence of stenosis and thrombosis of the fistula and the racial artery flow >=500 mL/min and the vein diameter >= 5 mm measured by duplex ultrasonography, or successful administration of hemodialysis with 2 needles with flow >= 350 mL/min.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando López Zárraga, Dr, Principal Investigator — Basque health System
Locations (1):
- Araba University Hospital (Santiago, Vitoria-Gasteiz, Spain